CLINICAL TRIAL: NCT04422444
Title: Characterization and Management of Post Intensive Care Syndrome in COVID19 Patients.
Brief Title: Post Intensive Care Syndrome in COVID19 Patients
Acronym: PICS-COVID19
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Sol Fernandez-Gonzalo, Postdoctoral neuropsychology researcher, Corporacion Parc Tauli
Other Study IDs: 2020/577
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: COVID19; Post Intensive Care Unit Syndrome
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Questionnaires — Participants will answer questionnaires in three areas: physical/functional, emotional status and cognitive status

SUMMARY:
This project is based in the implementation of a combined monitoring system (technological solutions and medical visits) in survivors of the critical illness due to the infectious disease by COVID-19. The main objective of the project is to characterize the Post-Intensive Care Syndrome (PICS) and detect early needs for specific treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU for COVID 19

Exclusion Criteria:

* Mental health diagnosis previous to the COVID19 infection
* Acquired brain damage or neurological disease previous to the COVID19 infection

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ICU patients with COVID19
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Short Form 12 Health Survey (SF12) at 12 month | Every month during a 12 months follow-up period
  Health related quality of live scale. Values are directly transformed in T scores (mean=50; SD=10), with higher scores meaning better outcome.

SECONDARY OUTCOMES:
Change from baseline Lawton & Brody Instrumental activities of daily living scale at 12 months | Every month during a 12 months follow-up period
  Measure of independent living skills. Values are from 0 to 8, with higher scores meaning better outcome.
Change from baseline Perceived Deficits Questionnaire (PDQ) at 12 months | Every month during a 12 months follow-up period
  Self-report measure of cognitive dysfunction. Values are from 0 to 22, with lower scores meaning better outcome.
Change from baseline Hospital Anxiety and Depression Scale (HADS) at 12 months | Every month during a 12 months follow-up period
  A self-assessment instrument for detecting states of depression and anxiety in the setting of an hospital medical outpatient. Values are from 0 to 42, with lower scores meaning better outcome.
Change from baseline Davidson Trauma Scale (DTS) at 12 months | Every month during a 12 months follow-up period. Values are from 0 to 136, with lower scores meaning better outcome.
  Self-report measure of Post Traumatic Stress Disorder (PTSD) symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: SOL FERNANDEZ, PhD, Principal Investigator — Institut d'Investigació i Innovació Parc Taulí (I3PT)
Locations (1):
- Corporació Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Fernandez-Gonzalo S, Navarra-Ventura G, Goma G, Godoy-Gonzalez M, Oliveras L, Ridao Sais N, Espinal C, Fortia C, De Haro C, Ochagavia A, Jodar M, Forne C, Santos-Pulpon V, Sarlabous L, Bacardit N, Subira C, Fernandez R, Palao D, Roca O, Blanch L, Lopez-Aguilar J. Characterization of postintensive care syndrome in a prospective cohort of survivors of COVID-19 critical illness: a 12-month follow-up study. Can J Anaesth. 2024 Sep;71(9):1282-1301. doi: 10.1007/s12630-024-02811-4. Epub 2024 Sep 9. PMID 39251486
- [Derived] Navarra-Ventura G, Godoy-Gonzalez M, Goma G, Jodar M, Sarlabous L, Santos-Pulpon V, Xifra-Porxas A, de Haro C, Roca O, Blanch L, Lopez-Aguilar J, Fernandez-Gonzalo S. Occurrence, co-occurrence and persistence of symptoms of depression and post-traumatic stress disorder in survivors of COVID-19 critical illness. Eur J Psychotraumatol. 2024;15(1):2363654. doi: 10.1080/20008066.2024.2363654. Epub 2024 Jun 17. PMID 38881386
- [Derived] Godoy-Gonzalez M, Navarra-Ventura G, Goma G, de Haro C, Espinal C, Fortia C, Ridao N, Miguel Rebanal N, Oliveras-Furriols L, Subira C, Jodar M, Santos-Pulpon V, Sarlabous L, Fernandez R, Ochagavia A, Blanch L, Roca O, Lopez-Aguilar J, Fernandez-Gonzalo S. Objective and subjective cognition in survivors of COVID-19 one year after ICU discharge: the role of demographic, clinical, and emotional factors. Crit Care. 2023 May 15;27(1):188. doi: 10.1186/s13054-023-04478-7. PMID 37189173